CLINICAL TRIAL: NCT04624646
Title: Clinical Implication of Atrial Fibrillation Detection Using Wearable Device in Patients With Cryptogenic Stroke - The Comparison Between Short-term Continuous Patch and Long-term Discontinuous Monitoring
Brief Title: Clinical Implication of Atrial Fibrillation Detection Using Wearable Device in Patients With Cryptogenic Stroke
Acronym: CANDLE-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CANDLE-AF Trial
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation; Ischemic Stroke; Transient Ischemic Attack
Keywords: Atrial fibrillation; Ischemic Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Ischemic Attack, Transient | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Conventional Holter Monitoring Group (Active Comparator): Holter monitoring is performed for 24 hours each at 1, 3, and 12 months after the diagnosis of stroke, and if atrial fibrillation is detected, the antiplatelet drug is changed to an anticoagulant.
  Interventions: Device: 24-hour Holter monitoring
- Discontinuous Monitoring Group (Experimental): Discontinuous ECG monitoring by finger contact is performed 3 times every day for 12 months after a stroke diagnosis. If atrial fibrillation is detected, the antiplatelet drug is changed to an anticoagulant.
  Interventions: Device: Discontinuous monitoring
- Single-lead Continuous Patch Group (Experimental): Continuous 72 hours of ECG monitoring by a single-lead patch is performed at a week and 1, 3, 6, 12 months after a stroke diagnosis. If atrial fibrillation is detected, the antiplatelet drug is changed to an anticoagulant.
  Interventions: Device: Continuous single-lead ECG Patch

INTERVENTIONS:
Device: Discontinuous monitoring — Discontinuous ECG monitoring by finger contact every day
  Arms: Discontinuous Monitoring Group
Device: Continuous single-lead ECG Patch — Continuous 72hr ECG monitoring by a single-lead patch at 3, 6, 9, 12 months after stroke
  Arms: Single-lead Continuous Patch Group
Device: 24-hour Holter monitoring — Continuous 24-hour monitoring by Holter monitor at 1, 6, 12 month after stroke
  Arms: Conventional Holter Monitoring Group

SUMMARY:
It is known that atrial fibrillation after stroke significantly increases the risk of stroke or systemic embolism. Accordingly, efforts have been made to detect hidden atrial fibrillation and apply treatment using anticoagulants instead of antiplatelet agents. The conventional method used to screen for atrial fibrillation in stroke patients who did not have atrial fibrillation at first admission is 24-hour Holter monitoring. This study will compare the detection rate of atrial fibrillation with discontinuous ECG monitoring three times a day and 72 hours of single-lead ECG patch monitoring compared with the conventional Holter test.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed brain infarction
* No history and diagnosis of atrial fibrillation at the time of admission
* Rejected implantable loop recorder
* Informed consent

Exclusion Criteria:

* Cannot use KardiaMobile system alone or with the help of others

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-09-18 (Estimated); Study Completion 2025-09-18 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation detection rate | Until 1 year after stroke
  Compare detection rates of each arms

SECONDARY OUTCOMES:
Recurrent stroke | Until 1 year after stroke
  Recurrent stroke
Major adverse cardiac and cerebrovascular event | Until 1 year after stroke
  composite of nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Junbeom Park, M.D., PhD., Principal Investigator — Ewha Womans University Mokdong Hospital; Tae-Jin Song, MD, Principal Investigator — Ewha Womans University Seoul Hospital; Dong-Hyeok Kim, MD, Principal Investigator — Ewha Womans University Seoul Hospital
Locations (9):
- South Korea (9):
  - Yonsei University Health System, Yongin Severance Hospital, Yongin, Gyeonggi-do
  - Ewha Womans University Seoul Hospital, Gangseo, Seoul
  - Hanyang University Seoul Hospital, Seongdong, Seoul
  - Ewha Womans University Mokdong Hospital, Yangcheon, Seoul
  - Daegu Catholic University Medical Center, Daegu
  - Gachon University Gil Hospital, Incheon
  - Kyung Hee University Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul